CLINICAL TRIAL: NCT04152902
Title: Quality of Life After Surgery for End-stage Achalasia: Pull-down Heller-Dor vs Esophagectomy
Brief Title: Quality of Life After Surgery for End-stage Achalasia
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Sandro Mattioli, Professor, University of Bologna
Other Study IDs: ESA
Record Dates: First submitted 2019-10-19; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Symptoms and Signs; Quality of Life
MeSH Terms: conditions — Signs and Symptoms | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 70 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PULL-DOWN HELLER-DOR: The PD-HD procedure aimed to restore the vertical axis of the intraabdominal portion of the oesophagus as much as possible. In brief, before performing the myotomy and the anterior fundoplication according to Dor, at least 6 cm of the mediastinal oesophagus was fully isolated; two or more U intramuscular stitches were applied on the curling of the right side of the oesophagus, pulled down and rotated towards the right side of the gastro-oesophageal junction. The PD-HD operation was performed under manometric control
  Interventions: Other: Objective outcome; Other: Quality of life
- OESOPHAGECTOMY: OE was performed with open technique, or recently, with a minimally invasive technique. The stomach was always the oesophageal substitute, and the oesophagogastric anastomosis was preferably located at the thoracic dome or at the neck to minimize the risk of postoperative reflux oesophagitis or cancer growth in the residual dilated oesophagus
  Interventions: Other: Objective outcome; Other: Quality of life

INTERVENTIONS:
Other: Objective outcome — The final outcome of surgical therapy was assessed according to a semi-quantitative scale graded as excellent, good, fair and poor, according to quantitative grades for dysphagia, reflux symptoms and oesophagitis
Other: Quality of life — SF-36 Questionnaire

SUMMARY:
Therapy for end-stage achalasia is under debate: comparative data on the long-term functional results of myotomy and oesophagectomy are lacking. The study aimed to compare the objective outcomes and quality of life after oesophageal myotomy and oesophagectomy.

The study included 31 patients (57 years) who underwent the Heller-Dor procedure with verticalisation of the distal oesophagus (pull-down technique dedicated to sigmoid oesophagus treatment) and 29 patients (recurrence free, 64 years) (p=0.539) who underwent oesophagectomy for end-stage achalasia or for cancer, extracted from a database designed for prospective clinical research. The objective outcomes of treatment were evaluated with semi-quantitative scales investigating dysphagia, reflux symptoms and endoscopic oesophagitis. Quality of life was assessed with the SF-36 questionnaire.

DETAILED DESCRIPTION:
Patients were extracted from a database designed for prospective clinical research on benign and malignant oesophageal diseases. For this study, the investigators considered patients who underwent operations for end-stage achalasia from January 1987-July 2018 and patients who survived after primary esophagectomy for oesophageal cancer between January 2008 and December 2018 without undergoing neoadjuvant/adjuvant therapy. End-stage achalasia was diagnosed on the basis of clinical history, upper gastrointestinal tract endoscopy and barium swallow results (oesophageal diameter larger than 6 cm, distal oesophagus kinked towards the left side, outside the axis). Standard oesophageal manometry, or more recently, high-resolution manometry, was routinely performed. Cases of pseudo-achalasia (oesophageal dilation secondary to organic stenosis of the cardia) were excluded based on clinical, endoscopic and histology patterns. In the presence of end-stage achalasia Pull-down Heller-Dor was the first primary treatment option for patients with the following: a) no severe mucosal inflammation or moderate/high grade dysplasia and b) redo surgery exclusively for dysphagia relapse due to insufficient myotomy. Esophagectomy was the treatment of choice for patients with the following: a) relapsed dysphagia after myotomy due to scarring that caused stenosis of the cardia, b) iterative surgery, c) cancerization risk patterns, and d) a diagnosis of cancer.

The pull-down Helle-Dor procedure aimed to restore the vertical axis of the intraabdominal portion of the oesophagus as much as possible. In brief, before performing the myotomy and the anterior fundoplication, at least 6 cm of the mediastinal oesophagus was fully isolated; two or more U intramuscular stitches were applied on the curling of the right side of the oesophagus, pulled down and rotated towards the right side of the gastro-oesophageal junction. The pull-down Heller-Dor operation was performed under manometric control.

Esophagectomy was performed with open technique, or recently, with a minimally invasive technique. The stomach was always the oesophageal substitute, and the oesophagogastric anastomosis was preferably located at the thoracic dome or at the neck to minimize the risk of postoperative reflux oesophagitis or cancer growth in the residual dilated oesophagus. Patients who underwent esophagectomy for cancer not related to achalasia were extracted from the relative case series to form a control group that matched the end-stage achalasia study group according to age and surgical technique; these patients had not undergone neoadjuvant or adjuvant chemotherapy and were cancer free at follow-up.

The duration of achalasia symptoms was calculated starting from the date of onset to the date of surgery at the investigator's institution. After surgery, the patients underwent a timed follow-up composed of clinical interviews, upper GI tract barium swallow and endoscopy. The symptoms were evaluated according to semi-quantitative scales graded from 0 (absence) to 3 (maximal intensity) based on Van Trappen's criteria for dysphagia and Visick's criteria for gastro-oesophageal reflux. Upper GI endoscopy aimed to detect post Heller's myotomy reflux oesophagitis, Barrett's oesophagus and areas suspected for dysplasia or cancer. Reflux oesophagitis was initially assessed according to the Savary-Miller and Ismail Beigi criteria and successively assessed according to the Los Angeles classification. The final outcome of surgical therapy was assessed according to a semi-quantitative scale graded as excellent, good, fair and poor, according to quantitative grades for dysphagia, reflux symptoms and oesophagitis.

Quality of life was assessed by the version of the 36-Item Short Form Survey (SF-36) validated for Italy. The questionnaire was a generic Health-Related Quality of Life (HRQL) measure that investigated eight specific health domains: physical functioning (PF), restrictions in activities due to physical (RP) or emotional health (RE), bodily pain (BP), general health (GH), vitality (VT), mental health (MH) and social functioning (SF). The SF-36 scores for each health domain ranged from 0 (poor HRQL) to 100 (best HRQL). Patients self-administered the questionnaires they received in mail for the specific purpose of this study.

ELIGIBILITY:
Inclusion Criteria patients with:

* follow-up longer than 1 year
* preoperative and postoperative endoscopy available
* preoperative and postoperative barium swallow available
* preoperative and postoperative manometry available

Exclusion criteria:

* patients undergone chemotherapy
* patients with relapse of disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Tertiary referral center
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 1987-01 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
change of dysphagia severity from preoperative to 3 years after surgery | 3 years
  changing of dysphagia severity from preoperative to 3 years after surgery. Dysphagia severity is evaluted according to a semiquantitative scale graded from 0 (absence) to 3 ( maximal intensity) based on Van Trappen's criteria
change of gastroesphageal reflux symptoms from preoperative to 3 years after surgey | 3 years
  change of gastroesphageal reflux symptoms from preoperative to 3 years after surgey. Severity of reflux symptoms was evaluated according to a semiquantitative scale graded from 0 (absence) to 3 ( maximal intensity) based on Van Trappen's criteria
change quality of life from preoperative to 3 years after surgery | 3 years
  change quality of life from preoperative to 3 years after surgery. The SF-36 questionnaire investigated eight specific health domains: physical functioning (PF), restrictions in activities due to physical (RP) or emotional health (RE), bodily pain (BP), general health (GH), vitality (VT), mental health (MH) and social functioning (SF). The SF-36 scores for each health domain ranged from 0 (poorer HRQL) to 100 (best HRQL).

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Thoracic Surgery Maria Cecilia Hospital, Cotignola, RA, Italy

IPD SHARING:
Plan to Share IPD: No